CLINICAL TRIAL: NCT04859959
Title: Gallium-68 Labeled Pentixafor PET/CT in the Diagnosis and Characterization of Adrenal Masses
Brief Title: Gallium-68 Labeled Pentixafor PET/CT in Adrenal Masses
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PenAM
Record Dates: First submitted 2021-04-22; First posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2020-07

CONDITIONS: Adrenal Mass

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-Pentixafor PET/CT scan (Experimental): Intravenous Inject 68Ga-Pentixafor and perform PET/CT scan 1h later.
  Interventions: Diagnostic Test: Gallium-68 Pentixafor PET/CT

INTERVENTIONS:
Diagnostic Test: Gallium-68 Pentixafor PET/CT — Intravenous injection of one dosage of 74-222 MBq (2-6 mCi) Gallium-68 Pentixafor. Tracer doses of Gallium-68 Pentixafor will be used to image adrenal lesions by PET/CT.

SUMMARY:
The CXC chemokine receptor type 4 (CXCR4), which is a G protein-coupled receptor expressed on the surface of the cell membrane, contributes to the development and progression of malignancies and functional endocrine disorders. CXCR4 expression has been reported to be upregulated in aldosterone-producing adenomas and cortisol-producing adenomas; however, its expression is almost negligible in non-functioning adrenal adenomas. Besides, CXCR4 is also hardly expressed by the tumor cells in paragangliomas. 68Ga-pentixafor, a CXCR4-specific PET tracer, may therefore be effective for the evaluation of the functional lateralization of adrenal lesion and identification of functional adrenocortical adenomas. In this pilot study, we aimed to develop 68Ga-pentixafor PET/CT as a noninvasive test for the recognition of functional adrenocortical lesions and to help guide the management of patients with suspicious adrenal masses.

DETAILED DESCRIPTION:
Identifying the functional distinctions between adrenal nodules remains challenging. It is imperative to employ the least invasive approach for the functional evaluation of adrenal masses (e.g., adrenal venous sampling) without compromising efficacy. The conventional functional diagnosis protocol of adrenal masses is based on a combination of clinical symptoms, the presence of adrenal hormonal disorders, and radiographic features. However, the clinical manifestations of endocrine diseases are diverse, and a lack of uniformity in diagnostic protocols and assay methods for determining hormonal activation in adrenal disorders results in a significant variability in measurements. Besides, conventional imaging provides information of the morphology of a lesion, but not its functional status. Thus, an effective and non-invasive workup is needed for the characterization of adrenal masses and their therapeutic management.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Patients with adrenal diseases.
* A diagnostic computed tomography (CT) or magnetic resonance imaging (MRI) of the adrenal region within the previous 6 months prior to dosing day is available

Exclusion Criteria:

* Pregnant or breast-feeding women.
* Prior or planned administration of a radiopharmaceutical within 8 half-lives of the radionuclide used on such radiopharmaceutical including at any time during the current study.
* Any mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study, and/or evidence of an uncooperative attitude

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
The diagnosis efficiency | through study completion, an average of 2 year
  The diagnosis efficiency of functional lateralization and identification of functional adrenocortical adenomas

SECONDARY OUTCOMES:
Standard uptake value (SUV) | From right after tracer injection to 2-hours post-injection
  Determination of SUV for detected lesions and normal liver and adrenal tissue of 68Ga-Pentixafor

CONTACTS AND LOCATIONS:
Overall Officials: Li Huo, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ding J, Li X, Liu S, Gao Y, Zheng G, Hacker M, Zhang Y, Tong A, Huo L. Clinical Value of 68Ga-Pentixafor PET/CT in Subtype Diagnosis of Primary Aldosteronism Patients with Adrenal Micronodules. J Nucl Med. 2024 Jan 2;65(1):117-124. doi: 10.2967/jnumed.123.266061. PMID 38050127